CLINICAL TRIAL: NCT06536101
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GIM-407 in Healthy Adult Participants
Brief Title: The Purpose of the Study is to Evaluate the Safety, Tolerability and Pharmacokinetics of Single-ascending and Multiple-ascending Doses of GIM-407
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgiamune Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GIM407-CT01
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: A first in human, randomized, double-blind, placebo-controlled, dose escalation study of single and multiple oral doses of GIM-407 in healthy adult participants. The study will include 3 parts, a single ascending dose (SAD) part (Part 1) and a multiple ascending dose (MAD) part (Part 2), and optional Food-effect cohorts (Part 3), which will proceed in a staggered manner with a partial overlap.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIM-407 oral dose (Experimental): SAD: Up to 5 ascending cohorts of subjects are planned to be orally dosed
  MAD: Up to 4 ascending dose cohorts of subjects are planned to be orally dosed once daily for 7 consecutive days
  Interventions: Drug: GIM-407
- Matching placebo oral dose (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GIM-407 — GIM-407 oral dose
  Arms: GIM-407 oral dose
Drug: Placebo — Matching placebo oral dose
  Arms: Matching placebo oral dose

SUMMARY:
This study is for the evaluation of the safety, tolerability, PK, PD, and biomarker activity of GIM-407 in healthy volunteers in the absence of any disease-related or potentially confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects (non childbearing or agree to use appropriate effective birth control),
* Nonsmoker or occasional smoker (ie, who smokes ≤10 cigarettes or equivalent of tobacco or nicotine-containing products, including vapes) per week within 30 days prior to Screening and is able to abide by the smoking policy of the study site during the in house observation period.

Exclusion Criteria:

* History or presence of any disease that affects drug absorption, distribution, metabolism, or excretion such as gastrointestinal dysfunction, peptic ulcer, gastrointestinal surgery, cholecystectomy, etc
* Any current active infections, including localized infections, or any recent history of active infections, cough, or fever within 1 week prior to study drug
* Known history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
* Use of any prescribed or nonprescribed medication (including over-the-counter medications, vitamins, multivitamins, recreational drugs, dietary supplements, and herbal remedies such as St. John's Wort extract) or drugs considered likely to interfere with the safe conduct of the study within 7 days or 5 half lives of the drug (whichever is longer) prior to the first dose
* Receipt of an investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non investigational intervention (drug, vaccine, or invasive medical device)
* Have received any live vaccines (bacterial or viral) within 30 days prior to the first dose of IP or intend to receive a live vaccine during the study period.
* Pregnant or breastfeeding female participant. Female participant who is planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety | Baseline through Study Completion (up to Day 14)
  Incidence of treatment emergent AEs
Evaluation of Safety | Baseline through Study Completion (up to Day 14)
  Change in laboratory safety assessments from baseline
Evaluation of Safety | Baseline through Study Completion (up to Day 14)
  Number of participants with clinically significant abnormal 12-lead ECG results as assessed by the investigator
Evaluation of Safety | Baseline through Study Completion (up to Day 14)
  Number of participants with abnormal physical examination findings as assessed by the investigator

SECONDARY OUTCOMES:
Area Under the Curve (AUC) will be assessed | Multiple timepoints from Baseline through Study Completion (up to Day 14)
  Area under the plasma concentration versus time curve
Maximum Blood Concentration (Cmax) will be assessed | Multiple timepoints from Baseline through Study Completion (up to Day 14)
  Maximum observed concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia